CLINICAL TRIAL: NCT04671901
Title: A Single Arm Open-Label Pilot Study of Prophylactic Romiplostim Use Compared to Benchmark Rate in the Prevention of Chemotherapy Induced Thrombocytopenia in Pediatric Solid Tumors Patients Undergoing Myelosuppressive Chemotherapy
Brief Title: A Study of Romiplostim to Prevent Low Platelet Counts in Children and Young Adults Receiving Chemotherapy for Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-467
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2023-03

CONDITIONS: Solid Tumor; Solid Tumor, Childhood; Solid Carcinoma
Keywords: romiplostim; primary solid tumor; Solid tumor; Solid tumor, childhood; Childhood solid tumor; Pediatric Solid Tumors; 20-467; Memorial Sloan Kettering Cancer Center
MeSH Terms: interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pediatric Participants (Experimental): Male and female patients aged 1-21 years with a primary solid tumor undergoing treatment with the pre-defined chemotherapy regimens of EFT, MAP or D9803.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Participants will receive weekly doses of romiplostim, beginning with cycle 4. The initial romiplostim dose will be 10 mcg/kg, and subsequent doses w ill vary based on chemotherapy regimen for a target of platelet count > 75,000- 200,000/mcL. Participants will continue romiplostim until completion of MAP or D9803, as defined above. Maximum romiplostim dose is 10 mcg/kg. Participants will be followed until 6 months after the last dose of romiplostim.

SUMMARY:
The purpose of this study is to find out whether romiplostim can help prevent low platelet counts caused by N8 or EFT chemotherapy, reduce the number of platelet transfusions required during chemotherapy, and prevent treatment delays due to low platelet counts.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of a primary solid tumor. Patients must have histological verification of malignancy at MSKCC.
* Male and female patients aged 1-21 years with a primary solid tumor undergoing treatment with the pre-defined chemotherapy regimens of EFT, MAP, D9803. Prior to enrollment patient could have been undergoing induction therapy with a similarly myelosuppressive regimen as long as they will be continuing with EFT, MAP, D9803 at the time of study enrollment.
* Patients undergoing treatment with MAP chemotherapy w ho have had ≥ 1 platelet transfusion during induction stage of treatment.
* Total Bilirubin (sum of conjugated + unconjugated) ≤ 3 times institutional upper limit of normal (ULN) for age and ALT/AST ≤ 3 times institutional ULN for age.
* Normal cardiac function:

  * Shortening fraction greater than or equal to 28% by echocardiogram OR Left ventricular ejection fraction (LVEF) greater than or equal to 50% on technetium- 99m pertechnetate radionuclide cineangiography (MUGA) or echocardiogram.
  * Screening ECG with corrected QT (QTc) interval of < 470 msec.
  * Timing of cardiac assessment: We will utilize the most recent EKG/ECHO when assessing cardiac function. See section 9.0 for additional details.
* Adequate renal function, defined as an estimated Creatinine Clearance or GFR >40ml/min or an normal creatine for age (see below)

Serum Creatinine by age:

Age (years) <6: Maximum Serum Creatinine (mg/dL), Male 0.8, Female 0.8 Age (years) 6 to <10: Maximum Serum Creatinine (mg/dL), Male 1, Female 1 Age (years) 10 to <13: Maximum Serum Creatinine (mg/dL), Male 1.2, Female 1.2 Age (years) 13 to <16: Maximum Serum Creatinine (mg/dL), Male 1.5, Female 1.4 Age (years) >16: Maximum Serum Creatinine (mg/dL), Male 1.7, Female 1.4

These threshold creatine values were derived from the Scwartz formula estimating GFR, utilizing child length and statured published by the CDC.

Exclusion Criteria:

* Patients with history of hematologic malignancies or allogenic/autogenic stem cell transplant.
* Patients with a currently known predisposition to a myeloid stem cell disorder, myeloid leukemia, and/or bone marrow failure syndrome including, but not limited to:

  * Aplastic anemia
  * Ataxia telangiectasia
  * Bloom syndrome
  * Congenital amegakaryocytic thrombocytopenia
  * Cyclic neutropenia
  * Diamond Blackfan anemia
  * Dyskeratosis congenita
  * Familial AML/MDS syndromes (including ANKRD26, CEBPA, DDX41, ETV6, GATA2, RUNX1, SRP72)
  * Fanconi anemia
  * Kostmann disease
  * Li-Fraumeni syndrome
  * Neurofibromatosis
  * Nijmegen breakage syndrome
  * Noonan syndrome
  * Paroxysmal nocturnal hemoglobinuria
  * Pearson syndrome
  * Poland syndrome
  * Rothmund-Thomson syndrome
  * Severe congenital neutropenia
  * Thrombocytopenia absent radii syndrome
  * Trisomy 8
  * Trisomy 21
  * WHIM syndrome
  * Wiskott Aldrich syndrome
  * Xeroderma pigmentosa
* Secondary malignancy in the past 5 years.
* Patients who have previously undergone up-front chemotherapy and have relapsed or progressed through therapy.
* Patients who have received 4 or more cycles of induction chemotherapy for their current malignancy prior to time of enrollment.
* Previous use of romiplostim, eltrombopag, recombinant human TPO, or any other TPO receptor agonist, or any investigational platelet producing agent.
* Patients receiving other investigational agents are not eligible for study entry.

History of uncontrolled arrhythmias, clinically significant electrocardiogram (ECG) abnormalities, active heart failure or pericardial disease.

* Patients with current or prior venous thrombotic event or arterial thrombotic event at time of enrollment will be ineligible for this study.
* Pregnant women/lactating mothers.
* Patients unwilling to use effective contraception method, which includes abstinence.
* Patients with an inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy.

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Ortiz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pediatric Participants
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pediatric Participants
Number analyzed (Participants) | 2
Age, Continuous [Median (Full Range); unit: years] | 14 [11 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Platelet Transfusions During the Studied Portions of the EFT or D9803 Cycles
Description: The primary purpose of this study is to evaluate whether romiplostim administration can decrease the total number of platelet transfusions required during the treatment courses of EFT or D9803 when compared to the benchmark rate.
Time Frame: up to 6 months
Population: N/A - data were not collected
Arm/Group | Pediatric Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Pediatric Participants
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT04671901/Prot_SAP_000.pdf